CLINICAL TRIAL: NCT04601311
Title: A Digitally Supported Guided Self-determination Intervention Versus Attention Control for People With Type 2 Diabetes in Outpatient Clinics - a Randomised Clinical Trial
Brief Title: A Guided Self-determination Intervention Versus Attention Control for People With Type 2 Diabetes in Outpatient Clinics
Acronym: OVERCOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Zoffmann, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P-2020-864
Record Dates: First submitted 2020-10-07; First posted 2020-10-23 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and treatment providers will not be blinded to the allocated trial intervention. The treatment providers are not involved in the analyses. All other medical personnel will be blinded by blinding of notes in the participant's electronic records. Outcome assessors and external statisticians at the Copenhagen Trial Unit will be blinded to the randomisation status of the participants. The statistical analyses will be conducted with the intervention groups coded as X and Y. The steering committee will write two abstracts while the blinding is intact, one assuming the experimental intervention group is X and the control intervention group is Y, and one assuming the opposite. After this, the code will be broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided self-determination (Experimental): 3 to 5 one-hour digital or analogue guided self-determination sessions
  Interventions: Behavioral: Guided self-determination
- Personal support in goal-pursuing (Active Comparator): Up to five personal goal pursuing support sessions
  Interventions: Behavioral: Personal support in goal-pursuing

INTERVENTIONS:
Behavioral: Guided self-determination — Before randomisation, the participants are supported in formulating one personal value-clarifying goal: 'One thing I want to achieve in my life with diabetes within a year is'….
  The goal is registered.
  Patients go through a guided self-determination intervention preparing themselves by completing reflection sheets, analogue or digital by patient's choice, and individually facilitated by a guided self-determination-certified nurse, face-to-face, over video or over telephone. Sessions scheduled every second week. Number of sessions 3-5 is decided at session 2.
  A relative may take part in one session completing an analogue reflection sheet as preparation.
  Participants continue usual care.
  Arms: Guided self-determination
Behavioral: Personal support in goal-pursuing — Before randomisation, the participants are supported in formulating one personal value-clarifying goal: 'One thing I want to achieve in my life with diabetes within a year is'….
  The goal is registered.
  Patients receive personal goal pursuing support up to five sessions, lasting up to one hour with a communication trained healthcare professional following up on the goal, face-to-face, digitally, or over telephone. The sessions are scheduled every second week. A relative may take part in one session.
  Participants continue usual care.
  Arms: Personal support in goal-pursuing

SUMMARY:
Background In management of type 2 diabetes, autonomy supporting interventions may be a prerequisite to achieve 'real life' patient engagement and more long-term improvement. Preliminary evidence has previously shown that the autonomy supporting intervention, guided self-determination method might have effect on HbA1c and diabetes distress in people with type 1 diabetes. However, previous trials were all rated as high risk of bias and did not assess potential harm of the the intervention. Thus, in the current trial, the objective is to investigate the benefits and harms of guided self-determination interventions versus an attention control group intervention in adults with type 2 diabetes.

Methods/design The trial planned is a randomised, pragmatic, investigator-initiated, dual-centre, parallel group, clinical superiority trial of guided self-determination intervention versus an attention control group for people diagnosed with type 2 diabetes in outpatient clinics. The participants (n=224) will be recruited from the department of Endocrinology at a University hospital of Copenhagen, the Capital Region of Denmark and from Steno Diabetes Center Odense, University hospital in the Southern Region of Denmark. The experimental stepped-care intervention will consist of 3-5 analogue or digitally provided guided self-determination sessions lasting up to one hour with a guided self-determination facilitator. The attention control group will receive similar number of sessions lasting up to one hour with a communication trained healthcare professional provided face-to-face, digitally, or over telephone.This trial protocol is guided by the SPIRIT and CONSORT guidelines. Participants will be included if they have type 2 diabetes, > 18 years old, and, are not pregnant. Participants will be assessed before randomisation, at 5- and 12-months follow-up. The primary follow-up timepoint will be 12-months follow-up. The primary outcome will be diabetes distress. Secondary outcomes will be quality of life, depressive symptoms, and adverse events not considered serious. Exploratory outcome will be glycated haemoglobin, motivation, and serious adverse events. Data will be collected using REDCap. The analyses will be performed using the statistical programme Stata version 16.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age.
* Diagnosed with type 2 diabetes ≥ 3 months according to the International Classification System of Diseases (ICD-11.2-11.9) [43].
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Prior participation in GSD course(s) for the past two years
* Lack of signed of informed consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
diabetes distress | The Problem area in diabetes (PAID) will be measured at 12-months follow-up. A higher score on the scale (0-100) indicate higher diabetes distress
  Assessed by the validated 20-item scale of diabetes-related distress burden, Problem Areas in Diabetes (PAID)

SECONDARY OUTCOMES:
Depressive symptoms | Hospital anxiety and depression scale (HADS) will be measured at 12-months follow-up. A higher score on the scale (0-42) indicate higher anxiety and depression
  Assessed by the Hospital Anxiety and Depression Scale (HADS)
Generic Quality of life: SF-36 | SF-36 will be measured at baseline 12-months follow-up.
  Generic quality of life assessed by SF-36 The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The lower the score the more disability.
Adverse events not considered serious | 12-months follow-up
  Assessed by the Negative Effects questionnaire (NEQ-20) at 12-months follow-up. A higher score (0-80) indicate more adverse events related to the intervention.
diabetes distress | Problem areas in diabetes (PAID) will be measured at 5 months follow-up. A higher score on the scale (0-100) indicate higher diabetes distress
  Assessed by the validated 20-item scale of diabetes-related distress burden, Problem Areas in Diabetes (PAID)

OTHER OUTCOMES:
Type of motivation (autonomous/external), controlled (external) or resigned (amotivated) regarding diabetes self-care practices | Assessed at 12-months follow-up.Autonomous motivation indicated by higher treatment self-regulation Questionnaire (TSRQ)-scores on autonomy (8-56) or autonomy-index (autonomy (8-56) minus control(9-63) or lower TSRQ-scores on amotivation (4-28)
  Assessed by the Treatment self-regulation Questionnaire
HbA1c | Assessed at baseline and 12-months follow-up.
  Assessed from the participants' record. A higher value indicate poorer glycaemic control
Proportion of participants with one or more serious adverse events in the intervention period | 12-months follow-up
  Defined according to the ICH-GCP definition, as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolonging of existing hospitalization and resulted in persistent or significant disability or jeopardized the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Anne Sophie Mathiesen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the International Committee of Medical Journal Editors (ICMJE), a detailed data sharing plan is a requirement. We adhere to the requirements with the following statements: Depersonalised individual patient data will be made available to increase transparancy and use of data. Immediately following publication the Trial Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, Analytic Code will be made available through a link for anyone who wishes to a access data. There will be no end date for this access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication the Trial Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, Analytic Code will be made available through a link for anyone who wishes to a access data
Access Criteria: There will be no end date for this access.

REFERENCES:
- [Derived] Mathiesen AS, Zoffmann V, Lindschou J, Jakobsen JC, Gluud C, Olsen MH, Rasmussen B, Marqvorsen EHS, Rothmann MJ. Detailed statistical analysis plan for a guided self-determination intervention versus an attention control for outpatients with type 2 diabetes in the randomised OVERCOME trial. Trials. 2024 Nov 11;25(1):751. doi: 10.1186/s13063-024-08589-6. PMID 39523352
- [Derived] Mathiesen AS, Zoffmann V, Skytte TB, Jakobsen JC, Gluud C, Lindschou J, Rasmussen B, Marqvorsen E, Thomsen T, Rothmann M. Guided self-determination intervention versus attention control for people with type 2 diabetes in outpatient clinics: a protocol for a randomised clinical trial. BMJ Open. 2021 Dec 23;11(12):e047037. doi: 10.1136/bmjopen-2020-047037. PMID 34949603